CLINICAL TRIAL: NCT01850537
Title: Prospective Study To Assess The Safety and Efficacy of the PROW LIF Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NLT Spine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN0171
Record Dates: First submitted 2013-04-30; First posted 2013-05-09 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Degenerative Disc Disease
Keywords: DDD; PROW; FUSION; eSPIN; Cage; IBF; Discectomy; Lumbar Fusion; TLIF; MIS
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm study (Experimental): treatment of degenerative disc disease using the PROW LIF
  Interventions: Device: treatment of degenerative disc disease using the PROW LIF

INTERVENTIONS:
Device: treatment of degenerative disc disease using the PROW LIF — TLIF procedure for the treatment of degenerative disc disease using the PROW LIF procedure (system)
  Other Names: PROW LIF Procedure

SUMMARY:
This is a prospective, single-arm, open-label, non-randomized study. The aim of the study is to assess the safety and efficacy of the Prow LIF procedure in Transforaminal Lumbar Interbody Fusion (TLIF) procedures for the treatment of subjects with symptomatic degenerative disc disease (DDD).

DETAILED DESCRIPTION:
Primary endpoints:

* Safety: Incidence of device-related anticipated and unanticipated serious adverse events (SAE). However, ALL complications and adverse events (AE) will be monitored and recorded.
* Primary radiographic effectiveness outcome parameter: evaluations of fusion rate.

ELIGIBILITY:
Inclusion Criteria:main Inclusion Criteria

1. Male and female between 18-65 years of age (skeletally mature).
2. Subjects suffering from degenerative disc disease (DDD) accompanied by back pain with leg pain at a single level between L2 and S1 confirmed by history and radiographic studies and that are scheduled for a fusion operation. DDD is determined to be present if one or more of the following are noted:

   1. instability (defined as angulation ≥ 5° and/or translation ≥ 4mm on flexion/extension radiographs);
   2. osteophyte formation;
   3. decreased disc height;
   4. ligamentous thickening;
   5. disc degeneration/herniation; or
   6. facet joint degeneration.
3. A pre-op Oswestry Low Back Pain Disability Questionnaire (ODI) score of 35 % or more;
4. Be non-responsive to non-operative treatment for at least 6 months;

   -

Exclusion Criteria:

1. The Antero-Posterior (AP) diameter (at midline) of the involved level is <31mm.
2. Any previous spinal surgery at the involved level;
3. Spondylolisthesis > grade I;
4. Ankylosed segment at the affected level;
5. History or radiographic evidence of osteoporotic fractures in the spine;
6. Paraparesis;
7. Progressive neurologic conditions;

   -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Fusion rate | 24 months follow up
  Primary radiographic effectiveness outcome parameter: evaluations of fusion. Fusion will be evaluated at 6 months, 12 months and 24 months post-op using plain radiographs (AP, lateral and flexion/extension films) and at 24 months using CT scan as well

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Leitner, MD Dr., Principal Investigator — Head of the Spine surgery department, Meir Hospital
Locations (1):
- Spine Surgery Department, Meir Hospital, Israel, Kfar Saba, Israel

REFERENCES:
- See also: NLT SPINE website — http://www.nlt-spine.com